CLINICAL TRIAL: NCT02329210
Title: Clinical Registry Investigating Bardet-Biedl Syndrome
Acronym: CRIBBS
Status: Recruiting | Type: Observational
Sponsor: Marshfield Clinic Research Foundation (Other)
Responsible Party: Principal Investigator, Jeremy Pomeroy, PhD, Director, Clinical Research Center, Marshfield Clinic Research Foundation
Other Study IDs: HAW10113
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Bardet-Biedl Syndrome
MeSH Terms: conditions — Bardet-Biedl Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Bardet-Biedl Syndrome (BBS) is a rare genetic disorder associated with a vast array of symptoms. The features of BBS are highly variable, even between siblings, making long-term follow-up and centralization of information vital to better understanding this complex disease and designing effective treatments.

Marshfield Clinic has developed the Clinical Registry Investigating Bardet-Biedl Syndrome (CRIBBS) to gather comprehensive health information from patients diagnosed with BBS in a single repository. This information will be used to inform patients, families, and physicians about the complex features of BBS and will serve as a platform for researchers to develop effective and targeted treatment strategies for patients with BBS.

CRIBBS is a web-based, confidential database and the privacy of patients enrolled in the registry will always be respected. Information maintained in the database will be identifiable only by an assigned study identification number, not by name. The registry strictly complies with HIPAA regulations. CRIBBS participants may be contacted periodically with information regarding clinical trials or research studies, but participation is entirely voluntary.

CRIBBS will bring together complex genetic and clinical information from BBS patients to accelerate research into effective treatments, attract additional researchers, and make it easier for researchers to identify patients and find funding for innovative studies.

DETAILED DESCRIPTION:
The Clinical Registry Investigating Bardet-Biedl Syndrome (CRIBBS) is an international registry for individuals with a rare genetic disorder called Bardet-Biedl syndrome (BBS). The registry is sustained by private philanthropic funding sources. The primary objective of establishing and sustaining CRIBBS is to enable clinical natural history studies and therapeutic trials in individuals with BBS.

Participation in CRIBBS is open to individuals meeting diagnostic criteria for BBS and/or genetic confirmation of the condition. Identification and recruitment of members will be accomplished in two approaches. First, family support organizations will share information regarding CRIBBS and encourage enrollment in the registry. Second, a website will be developed for participants, families and health care providers. This website provides a portal for registration as well as medical and new information impacting health care for individuals with BBS.

Selection and Enrollment of Participants:

A website portal at www.bbs-registry.org facilitates voluntary registration of interested individuals. A CRIBBS coordinator will contact the individual and/or family to establish that participants meet published diagnostic criteria and/or genetic criteria for BBS. Individuals meeting criteria will be consented and assigned a unique identifier.

Data collection:

Consented participants and/or their parent/guardian will be interviewed by a CRIBBS coordinator to collect demographic information as well as completion of a health questionnaire. Because CRIBBS is an international study and participants are geographically dispersed most individuals will be interviewed using secured telephone or Internet services. Participants will also be asked to complete behavioral health surveys. Health information from providers and treatment facilities will be obtained with appropriate authorization. The CRIBBS coordinator will conduct an annual update of health information and the behavioral health surveys will be repeated.

Data Safety Monitoring:

* Participant confidentiality: Participation in CRIBBS is voluntary and every effort will be made to ensure participant privacy. Interviews with participants will be carried out by a CRIBBS coordinator in closed room. Personal Health Information obtained for health information abstraction will be stored securely in a double locked environment and destroyed following data abstraction. CRIBBS makes use primarily of an electronic database which is password protected and only accessible to CRIBBS staff members.
* Data use: Participant information will be used to inform researchers of the natural history of BBS, refine research initiatives and facilitate new therapies for individuals with BBS. De-identified data will be shared researchers and organizations approved by the CRIBBS board of directors.
* Registry Oversight: The Marshfield Clinic Research Foundation Institutional Review Board provides oversight of the CRIBBS registry while the CRIBBS board of directors determine the direction and focus of the registry.

ELIGIBILITY:
Inclusion Criteria: (1) Genetic confirmation of BBS or (2) manifest four primary features of BBS or (3) manifest three primary features plus two secondary features.

Primary Features: Rod-Cone dystrophy, Polydactyly, Obesity, Learning disabilities, Hypogonadism in males, Renal anomalies

Secondary Features: Speech disorder/delay, Strabismus/cataracts/astigmatism, Brachydactyly/syndactyly, Developmental delay, Polyuria/polydipsia, Ataxia/poor coordination/imbalance, Mild spasticity (especially lower extremities), Left ventricular hypertrophy/congenital heart disease, Hepatic fibrosis

Exclusion Criteria:

Individuals not meeting established genetic and/or phenotypic criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals meeting the diagnostic criteria of Bardet-Biedl syndrome and/or with genetic confirmation of the condition are eligible for participation in CRIBBS. Deceased individuals meeting diagnostic and/or genetic criteria may also be enrolled by their next of kin.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2014-06; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Registry Investigating Bardet-Biedl Syndrome | 15 years
  Natural history observational study of Bardet-Biedl syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Haws, M.D., Principal Investigator — Marshfield Clinic Research Institute
Locations (1):
- Marshfield Clinic Research Foundation, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haws RM, Kretz AD, Stankowski RV, Steiner RD. Bardet-Biedl syndrome: A model for translational research in rare disease. New Horizons in Translational Medicine 2: 102-109, 2015.
- [Background] Haws RM, Joshi A, Shah SA, Alkandari O, Turman MA. Renal transplantation in Bardet-Biedl Syndrome. Pediatr Nephrol. 2016 Nov;31(11):2153-61. doi: 10.1007/s00467-016-3415-4. Epub 2016 Jun 1. PMID 27245600
- [Background] Panny A, Glurich I, Haws RM, Acharya A. Oral and Craniofacial Anomalies of Bardet-Biedl Syndrome: Dental Management in the Context of a Rare Disease. J Dent Res. 2017 Nov;96(12):1361-1369. doi: 10.1177/0022034517716913. Epub 2017 Jun 29. PMID 28662344
- [Background] Olson AJ, Krentz AD, Finta KM, Okorie UC, Haws RM. Thoraco-Abdominal Abnormalities in Bardet-Biedl Syndrome: Situs Inversus and Heterotaxy. J Pediatr. 2019 Jan;204:31-37. doi: 10.1016/j.jpeds.2018.08.068. Epub 2018 Oct 4. PMID 30293640
- [Background] Pomeroy J, Krentz AD, Richardson JG, Berg RL, VanWormer JJ, Haws RM. Bardet-Biedl syndrome: Weight patterns and genetics in a rare obesity syndrome. Pediatr Obes. 2021 Feb;16(2):e12703. doi: 10.1111/ijpo.12703. Epub 2020 Jul 22. PMID 32700463
- [Background] Meyer JR, Krentz AD, Berg RL, Richardson JG, Pomeroy J, Hebbring SJ, Haws RM. Kidney failure in Bardet-Biedl syndrome. Clin Genet. 2022 Apr;101(4):429-441. doi: 10.1111/cge.14119. PMID 35112343